CLINICAL TRIAL: NCT04920253
Title: Real World Evidence with the Debritom+ TM Novel Micro Water Jet Technology At a Single Wound Center
Acronym: EVIDENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medaxis, LLC (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEDX-DT-03
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer; Surgical Wound Dehiscence; Traumatic Wounds
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Surgical Wound Dehiscence

STUDY DESIGN:
Intervention Model Description: Prospective, single-blinded, single-center, parallel group, randomized controlled trial (RCT). Control and Treatment Arms
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Prescribing Physician will be blinded. A site blinded physician will confirm the Prescribing Physician's initial assessment of wound healing and a final blinded Independent Adjudicator will review baseline and final images to assess and provide confirmation of healing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- debritom+ (Experimental): Group 1: Medaxis debritom+
  Interventions: Device: Study Device Debridement
- Sharp Scalpel (Active Comparator): Group 2: SOC (Sharp Scalpel Debridement)
  Interventions: Device: SOC Debridement

INTERVENTIONS:
Device: Study Device Debridement — debritom+ water jet debridement
  Arms: debritom+
Device: SOC Debridement — Sharp Scalpel
  Arms: Sharp Scalpel

SUMMARY:
Prospective, single-blinded, single-center, parallel group, randomized controlled trial (RCT) to assess rate and frequency of wound healing and associated financial savings, when using Medaxis debritom+ versus standard of care as a choice of debridement method, where both arms follow normal wound care practice in use of advanced wound care treatments.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to assess the clinical performance of the Medaxis debritom+ versus standard of care (sharp debridement using scalpel) in the real world practice of wound care management in a single center trial by collecting data on wound healing rates over time, success of advanced wound care treatments, and downstream financial costs in the treatment of diabetic foot ulcers, venous leg ulcers, dehisced surgical wounds and traumatic wounds. Medaxis debritom+TM is an advanced micro fluid jet FDA registered Class II device, which will be used within the cleared intended use of wound therapy.

ELIGIBILITY:
Inclusion Criteria:

General

Potential subjects are required to meet all of the following criteria for enrollment into the study and subsequent randomization:

1. At least 18 years old.
2. The index wound (i.e. current episode of the wound or ulceration) has been present for greater than 4 weeks prior to SV 1 and has had less than 1 year of documented medical treatment, as of the subject's consent for the study participation.
3. The index wound is a minimum of 1.0 cm2 and a maximum of 25 cm2 at SV1.
4. Subject understands and is willing to participate in the clinical study and can comply with weekly visits.
5. Subject must have read and signed the IRB approved Informed Consent Form (ICF) before study specific screening procedures that are not standard of care are undertaken.

   DFU
6. Presence of diabetic foot ulcer (DFU) that meets all of the following features:
7. Wagner Grade 1 or 2 (see Appendix A for definitions), including wounds that extend to the ligament, tendon, joint capsule or fascia
8. Without abscess or osteomyelitis
9. The index ulcer will be the largest ulcer if two or more DFUs are present and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2cm distant from index ulcer (edge to edge).
10. The index ulcer has been offloaded for at least 14 days prior to randomization
11. Adequate circulation to the affected foot as documented by a Clarifi SFDI Vascular Assessment Tool, or an Ankle Brachial Index (ABI) between 0.7 and 1.3 within 3 months of SV1, using the affected study extremity. As an alternative, arterial Doppler ultrasound can be performed, evaluating for bi-phasic dorsalis pedis and posterior tibial vessels at the level of the ankle within 3 months of SV1 or if monophasic wave forms present must have adequate micro circulation as evidenced by Clarifi SFDI Vascular Assessment Tool. Note: A documented record of an ABI test performed using the index ulcer leg, within 3 months of SV1 is acceptable for the purposes of this study. Otherwise, this must be completed in the Screening Visit. Acceptable alternatives include arterial Doppler ultrasound evaluating vessels at the level of the ankle, or documented adequate microcirculation as determined by a Clarifi SFDI Vascular Assessment Tool.

    VLU
12. All wounds using the CEAP VLU Classification, except for those in the exclusion criteria. (See Appendix A for definitions)
13. The index ulcer will be the largest ulcer if two or more VLUs are present and will be the only one evaluated in the study. If other Ulcerations are present on the same leg, they must be more than 2cm distant from index ulcer.
14. Adequate circulation to the affected foot as documented by a Clarifi SFDI Vascular Assessment Tool, or an Ankle Brachial Index (ABI) between 0.7 and 1.3 within 3 months of SV1, using the affected study extremity. As an alternative, arterial Doppler ultrasound can be performed, evaluating for bi-phasic dorsalis pedis and posterior tibial vessels at the level of the ankle within 3 months of SV1 or if monophasic wave forms present must have adequate micro circulation as evidenced by Clarifi SFDI Vascular Assessment Tool. Note: A documented record of an ABI test performed using the index ulcer leg, within 3 months of SV1 is acceptable for the purposes of this study. Otherwise, this must be completed in the Screening Visit. Acceptable alternatives include arterial Doppler ultrasound evaluating vessels at the level of the ankle, or documented adequate microcirculation as determined by a Clarifi SFDI Vascular Assessment Tool.

    Surgical Dehisced
15. All wounds using the Sandy Grading System, except those in the exclusion criteria. (See Appendix A for definitions)

    Traumatic
16. All wounds as per the CDC Surgical Wound Classification, with the exception of Class IV or dirty infected wounds, SSI - Deep incisional and organ space. (See Appendix A for definitions)

Exclusion Criteria:

General

Potential subjects meeting any of the following criteria will be excluded from enrollment and subsequent randomization:

1. The index wound, in the opinion of the investigator, is suspicious for cancer or have a positive carcinoma diagnosis.
2. Subject has a history of more than two weeks of treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the wound surface within 1 month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study.
3. Subject is taking a selective COX-2 inhibitor, such as Celecoxib, for any condition.
4. Subject is on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1.
5. History of radiation at the wound site (regardless of time since last radiation treatment).
6. Index wound has been previously treated or will need to be treated with any prohibited therapies (See Section 6 of this protocol for a list of prohibited medications and therapies).
7. Subject has a previous diagnosis of HIV, Hepatitis C, or other contagious diseases.
8. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or the subject has a known history of poor adherence with medical treatment.
9. Subject is pregnant or breast-feeding.
10. Presence of diabetes with poor metabolic control as documented with an HbA1c >12.0 % within 90 days of randomization.
11. Subject has end-stage renal disease as evidenced by a serum creatinine > 3.0mg/dL within 6 months of randomization.
12. BMI >55
13. PAR experiences a >30% change between SV1 and SV2 DFU
14. Wagner 2 wounds that require debridement of bone.
15. Osteomyelitis or bone infection of the affected foot as verified by x-ray, CAT Scan, or MRI within 30 days prior to randomization (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).

    VLU
16. Exclude

    1. Secondary post thrombotic
    2. Venous Obstruction
    3. Venous Obstruction with reflux
    4. Lipodermato sclerosis or atrophic blanche
17. Osteomyelitis or bone infection of the affected leg as verified by x-ray, CAT Scan, or MRI within 30 days prior to randomization (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).

    Surgical Dehisced
18. Using the Sandy Grading System for Surgical Wound Dehiscence: Wounds Grade 3 where organs are exposed, and 3a, where the infection is severe as deemed by the Principal Investigator.

    Traumatic
19. Using CDC Surgical Wound Classification, exclude

    1. Class IV - dirty infected wounds
    2. SSI - Deep incisional and organ space

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | 20 weeks
  Time to heal

SECONDARY OUTCOMES:
Complications | 20 weeks
  Incidence of all index wound-related complications (eg. cellulitis or Infection), hospitalization, wound recurrence
Advanced Wound Care Treatments | 20 weeks
  Number of successful advanced wound care treatments placed (eg. Negative Pressure Wound Therapy /grafts)
Cost | 20 weeks
  Cost of Treatment (including Advance Wound Care) and including any index wound-related, event-driven complications using patient records or Medicare reimbursement method.
Healed Proportion | 20 weeks
  Proportion of wounds completely healed

OTHER OUTCOMES:
Unhealed Proportion | 20 weeks
  Proportion of wounds not completely healed
PAR | 20 weeks
  Percent Area Reduction of Wound
AWC Failure | 20 weeks
  Number of failures in regard to advanced wound care treatments

CONTACTS AND LOCATIONS:
Overall Officials: Melvin B Price, DPM, Principal Investigator — MCR Health Inc.
Locations (1):
- MCR Health, Inc., Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No